CLINICAL TRIAL: NCT06158711
Title: A Retrospective Study of the Effect of Different Drugs Co-administration in the Treatment of Heart Failure
Brief Title: Real-world Research : Assessment of Effect of Combination of Drugs in the Treatment of Heart Failure
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Guang Yang, Director of Department of Gerontology/ Health Care and Medicine (Cardiology) , the First Affiliated Hospital of Shandong First Medical University &Shandong Provincial Qianfoshan Hospital, Qianfoshan Hospital
Other Study IDs: Qianfoshan HF 2023
Record Dates: First submitted 2023-11-16; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- single drug group, two drugs group, three drugs group and four drugs group: single drug group, patients with heart failure only took one sort of drugs two drugs group, patients with heart failure took two sorts of drugs three drugs group, patients with heart failure took three sorts of drugs four drugs group, patients with heart failure took four sorts of drugs

SUMMARY:
The goal of this observational study is to assess the effect of the different combination of drugs in the treatment of heart failure.

The main questions it aims to answer are:

* [question 1] The changes of BNP and LVEF in patients of each groups with different drugs co-administration.
* [question 2] The days of hospitalization, degree of lower limb edema (mild, moderate, severe) and 6-minute walking test in each groups.

Participants will be asked to do nothing. All the records of the patients will be download from the Big Data Cloud Platform of Health Care in the First Affiliated Hospital of Shandong First Medical University.

There is not a comparison group.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy and cost-effective of different drugs co-administration in the treatment of heart failure. For different reasons, patients with heart failure took different drug prescriptions. Now there are five kinds of drugs for the treatment of heart failure, such as angiotensin converting enzyme inhibitor or angiotensin receptor blocker (ACEI/ARB), beta-blokers, spironolactone, sodium-glucose cotransporter (sglt) 2 inhibitors and vericiguat. Our purpose is to assessment the efficacy and cost-effective of different drugs co-administration in the treatment of heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as "heart failure" or "cardiac insufficiency" on the first page of the medical record

Exclusion Criteria:

* Severe impairment of liver, kidney and lung function (transaminase increased more than 2 times; Scr > 265umol/L); malignant tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The hospitalized patients who were treated in the First Affiliated Hospital of Shandong First Medical School from January 2013.to October 2023
Sampling Method: Non-Probability Sample
Enrollment: 702 (Estimated)
Dates: Start 2023-11-30 (Estimated); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
The B-type natriuretic peptide (BNP) | Admission to hospital and 12 months thereafter
  B-type natriuretic peptide (BNP) is a marker of heart failure. Its levels can be measured with a rapid and commercially available bed-side assay. Rising levels correlate with the degree of left ventricular dysfunction and severity of symptoms.
Left ventricular ejection fraction (LVEF) of patients | Admission to hospital and 12 months thereafter
  Echocardiography is the gold standard for establishing the presence of left ventricular dysfunction. Left ventricular ejection fraction (LVEF) is the central measure of left ventricular systolic function. LVEF is the fraction of chamber volume ejected in systole (stroke volume) in relation to the volume of the blood in the ventricle at the end of diastole (end-diastolic volume).
Hospital mortality | Index hospital stay
  We recorded the death from heart failure, no matter the mode of death.

SECONDARY OUTCOMES:
Days of hospitalization and expenses of patients | Index hospital stay
  The hospitalization days and expenses of patients admitted with different drugs treatment were examined.
degree of lower limb edema (mild, moderate, severe) | Admission to hospital and 12 months thereafter
  Lower-extremity edema is one of the important factors in diagnosing, monitoring, and managing HF status. A senior cardiologist checked carefully for the presence of bilateral lower-extremity edema and graded its severity on a scale of 1 of 4 based on the extent of the edema in the leg, as follows: (1) none, (2) up to the height of the ankle level (mild edema), (3) up to the height of the knee (moderate edema), and (4) higher than knee level (severe edema).
6-minute walking test | Admission to hospital and 12 months thereafter
  The 6-minute walking test (6MWT) is a widely available and well-tolerated test for the assessment of the functional capacity of patients with HF.

CONTACTS AND LOCATIONS:
Overall Officials: Guang Yang, PhD, Principal Investigator — Qianfoshan Hospital

IPD SHARING:
Plan to Share IPD: Yes
patient characteristics and clinical outcomes
Supporting Information: Study Protocol, SAP
Time Frame: From 2024-8-1to 2027-8-1
Access Criteria: No criteria

REFERENCES:
- [Background] Kavalieratos D, Gelfman LP, Tycon LE, Riegel B, Bekelman DB, Ikejiani DZ, Goldstein N, Kimmel SE, Bakitas MA, Arnold RM. Palliative Care in Heart Failure: Rationale, Evidence, and Future Priorities. J Am Coll Cardiol. 2017 Oct 10;70(15):1919-1930. doi: 10.1016/j.jacc.2017.08.036. PMID 28982506
- [Background] Shen L, Claggett BL, Jhund PS, Abraham WT, Desai AS, Dickstein K, Gong J, Kober LV, Lefkowitz MP, Rouleau JL, Shi VC, Swedberg K, Zile MR, Solomon SD, McMurray JJV. Development and external validation of prognostic models to predict sudden and pump-failure death in patients with HFrEF from PARADIGM-HF and ATMOSPHERE. Clin Res Cardiol. 2021 Aug;110(8):1334-1349. doi: 10.1007/s00392-021-01888-x. Epub 2021 Jun 8. PMID 34101002
- [Background] Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Colvin MM, Drazner MH, Filippatos GS, Fonarow GC, Givertz MM, Hollenberg SM, Lindenfeld J, Masoudi FA, McBride PE, Peterson PN, Stevenson LW, Westlake C. 2017 ACC/AHA/HFSA Focused Update of the 2013 ACCF/AHA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Failure Society of America. J Am Coll Cardiol. 2017 Aug 8;70(6):776-803. doi: 10.1016/j.jacc.2017.04.025. Epub 2017 Apr 28. No abstract available. PMID 28461007
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; ESC Scientific Document Group. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC)Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2016 Jul 14;37(27):2129-2200. doi: 10.1093/eurheartj/ehw128. Epub 2016 May 20. No abstract available. PMID 27206819
- [Background] Vaduganathan M, Claggett BL, Jhund PS, Cunningham JW, Pedro Ferreira J, Zannad F, Packer M, Fonarow GC, McMurray JJV, Solomon SD. Estimating lifetime benefits of comprehensive disease-modifying pharmacological therapies in patients with heart failure with reduced ejection fraction: a comparative analysis of three randomised controlled trials. Lancet. 2020 Jul 11;396(10244):121-128. doi: 10.1016/S0140-6736(20)30748-0. Epub 2020 May 21. PMID 32446323
- [Background] Castiglione V, Aimo A, Vergaro G, Saccaro L, Passino C, Emdin M. Biomarkers for the diagnosis and management of heart failure. Heart Fail Rev. 2022 Mar;27(2):625-643. doi: 10.1007/s10741-021-10105-w. Epub 2021 Apr 14. PMID 33852110
- [Background] Authors/Task Force Members:; McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: Developed by the Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC). With the special contribution of the Heart Failure Association (HFA) of the ESC. Eur J Heart Fail. 2022 Jan;24(1):4-131. doi: 10.1002/ejhf.2333. PMID 35083827
- [Background] Heidenreich PA, Bozkurt B, Aguilar D, Allen LA, Byun JJ, Colvin MM, Deswal A, Drazner MH, Dunlay SM, Evers LR, Fang JC, Fedson SE, Fonarow GC, Hayek SS, Hernandez AF, Khazanie P, Kittleson MM, Lee CS, Link MS, Milano CA, Nnacheta LC, Sandhu AT, Stevenson LW, Vardeny O, Vest AR, Yancy CW. 2022 AHA/ACC/HFSA Guideline for the Management of Heart Failure: Executive Summary: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2022 May 3;145(18):e876-e894. doi: 10.1161/CIR.0000000000001062. Epub 2022 Apr 1. PMID 35363500
- [Background] Ji PJ, Zhang ZY, Yan Q, Cao HL, Zhao YJ, Yang B, Li J. The cardiovascular effects of SGLT2 inhibitors, RAS inhibitors, and ARN inhibitors in heart failure. ESC Heart Fail. 2023 Apr;10(2):1314-1325. doi: 10.1002/ehf2.14298. Epub 2023 Feb 1. PMID 36722326